CLINICAL TRIAL: NCT03099707
Title: The Treatment Ambassador Program: Pilot Testing a Peer-driven Intervention to Increase Treatment Initiation Among HIV-positive South Africans
Brief Title: The Treatment Ambassador Program: A Pilot Intervention to Increase Treatment Initiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Ingrid Theresa Katz, M.D., Assistant Professor and Research Scientist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P002222
Record Dates: First submitted 2017-03-17; First posted 2017-04-04 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-10

CONDITIONS: HIV
Keywords: Treatment; ART; South Africa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants are administered baseline, 3 month, and 6 month questionnaires and provided with study incentive (100 Rand per survey plus an additional 200 Rand to complete all three surveys) only. This group will not receive any additional engagement to care intervention. Investigators intend to follow their clinical outcomes through medical registries, pharmacy data, and the National Health Laboratory Service (a national database for all individuals living with HIV in South Africa regarding engagement in care).
- Treatment Ambassador Intervention (Active Comparator): Participants are administered baseline, 3 month, and 6 month questionnaires and provided with study incentive (100 Rand per survey plus an additional 200R to complete all three surveys). For participants randomized to the intervention arm, they will immediately meet with a Treatment Ambassador to begin the 8 session intervention, which has components of motivational interviewing, peer-support, and peer navigation. The protocol is detailed in a study manual that has been reviewed and undergone multiple iterative revisions to ensure cultural acceptability.
  Interventions: Behavioral: Treatment Ambassador

INTERVENTIONS:
Behavioral: Treatment Ambassador — This multi-component intervention, titled the "Treatment Ambassador Program," will target people living with HIV who have not initiated ART within 3 months of testing positive. Our intervention will last for 8 sessions over 8-14 weeks, and will aim to address the three steams of influences on decision-making through a system of patient navigation and support with an assigned partner living with HIV who is trained in motivational interviewing. It will be aimed at addressing barriers to ART initiation identified through our prior qualitative research, as framed through the Theory of Triadic Influence, by addressing the three streams of influences on decision-making through a system of patient navigation and support.
  Arms: Treatment Ambassador Intervention

SUMMARY:
This study will evaluate the feasibility and acceptability of the Treatment Ambassador program - a peer-supported intervention targeting individuals living with HIV who have not started on treatment within at least 3 months of testing.

DETAILED DESCRIPTION:
Global HIV treatment initiatives have focused on increasing access to antiretroviral therapy (ART), with the goal of creating an "AIDS-free generation." There is growing evidence, however, that treatment availability alone is insufficient to stop the spread of the disease. Countries where HIV is hyperendemic, such as South Africa, will not achieve population-level reductions in HIV until incident infections have been dramatically reduced over a lifetime, and people living with HIV (PLWH) no longer wait to start treatment until they have symptoms of advanced AIDS. As South Africa expands ART eligibility to all people living with HIV, it remains unclear if promoting earlier ART initiation will lead to widespread uptake. These operational realities raise two fundamental questions: how will we close the gap from the 3.4 million PLWH currently on ART to treating the over seven million people who need care; and what does this portend for the future of Treatment as Prevention in South Africa? The investigators' prior research suggests that optimizing ART initiation for PLWH in South Africa will require an intervention to reduce individual barriers to starting ART, promote social support, and enhance linkages to the healthcare system. In the proposed study, the investigators will build upon our prior research to pilot test a socio-behavioral multi-component peer intervention, to ensure that South Africans living with HIV initiate and sustain treatment. Investigators will test this intervention through a pilot randomized-controlled trial. This multi-component intervention is designed to address barriers to ART initiation identified in prior qualitative research, framed through the Theory of Triadic Influence (TTI). TTI focuses upon three "streams of influence" that impact health behavior at the individual-, social-, and structural-levels. The intervention will be delivered by "Treatment Ambassadors," who are PLWH who will function in multiple capacities, and have received intensive training in motivational interviewing (MI), peer-support, and peer navigation. They will then provide the intervention in eight sessions over 8-14 weeks. The intervention will be individually tailored to address the three streams of influence on patient decision-making as follows: MI will address individual perceived risk and ambivalence in decision-making; peer-support will target interpersonal social factors; and patient navigation will promote ART initiation and counter structural barriers.

Investigators will enroll 90 participants (45 in each arm) with the goal of assessing feasibility and acceptability. Investigators enrolled 84 participants in total. The 90 participant mark was not met due to time constraints and our eligibility requirements. In addition, preliminary efficacy will be assessed through the following measures:

Primary Outcome Measure: Timely ART initiation (initiation within 3 months of enrollment) (assessed through the National Health Laboratory Service, pharmacy records, and medical chart abstraction).

Secondary Outcomes Measures: 1) HIV-1 RNA Suppression within the first 6 months of study enrollment (assessed through the National Health Laboratory Service).

2) Behavioral Factors associated with failure to initiate ART in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

1. Adults living with HIV who are 18 years and older, who have not initiated ART within 3 months of learning their status
2. ART naïve,
3. Live within 60 km the testing center (due to prohibitive costs of following participants to remote locations);
4. English or Xhosa speaking; and
5. Eligible for treatment under current South Africa guidelines

Exclusion Criteria:

1. Unable to provide informed consent (e.g., due to intoxication or mental incapacity,
2. Persons less than 18 years of age,
3. Women who report current pregnancy at the time of consent. We are choosing to not include pregnant women in this study, because the study's recruitment site refers pregnant clients to more specialized care facilities that may better suit their needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Katz, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Desmond Tutu HIV Foundation, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Katz IT, Bogart LM, Fitzmaurice GM, Staggs VS, Gwadz MV, Bassett IV, Cross A, Courtney I, Tsolekile L, Panda R, Steck S, Bangsberg DR, Orrell C, Goggin K. The Treatment Ambassador Program: A Highly Acceptable and Feasible Community-Based Peer Intervention for South Africans Living with HIV Who Delay or Discontinue Antiretroviral Therapy. AIDS Behav. 2021 Apr;25(4):1129-1143. doi: 10.1007/s10461-020-03063-1. Epub 2020 Oct 30. PMID 33125587

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Started | 43 | 41
Completed | 43 | 37
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Treatment Ambassador Intervention | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 41 | 84
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [30 to 43] | 34 [21 to 48] | 34 [29 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 10 | 5 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 43 | 41 | 84
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 43 | 41 | 84

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Initiation at 3 Months After Study Enrollment
Description: Treatment Initiation will be measured at 3 months through clinic records, pharmacy data, and the National Health Laboratory Service (NHLS), a national database in South Africa. Primary data analysis will be an intent-to-treat analysis, which includes all randomized participants. Of note, every attempt will be made to continue assessing participants even if they drop out of treatment. In addition, investigators will replicate all analyses with the completers only. The hypothesis that the intervention will yield higher rates of antiretroviral therapy (ART) initiation by the completion of the intervention will be tested using Fisher's exact test; the treatment effect estimate will be summarized in terms of a relative risk and 95% confidence interval. Any baseline demographic or clinical variables identified as necessary covariates in preliminary analyses will be included in a logistic regression analysis that examines the main effect of treatment condition on the rates of ART initiation.
Time Frame: 3 months
Population: All participants who completed the full 6 months of the study were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 37
Participants | 1 | 5
Statistical Analysis 1: Comparison: Standard of Care vs Treatment Ambassador Intervention; Test type: Superiority; p = 0.105, Fisher Exact; Risk Ratio (RR) = 5.2, 95% CI 2-sided [0.6 to 43]

2. Secondary Outcome: HIV-1 RNA Suppression at 6 Months Post-enrollment
Description: HIV-1 RNA will be measured at 6 months year post enrollment among participants who start ART to allow for sub-group analyses of people living with HIV who start ART in the intervention vs. control groups. This will be accessible through NHLS and clinic data.
Time Frame: 6 months
Population: Data were not collected for participant HIV-1 RNA suppression at 6 months post-enrollment
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: CD4
Description: Mean CD4 counts at the 6 month assessment
Time Frame: 6 months
Population: No CD4 data were collected at 6 months
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Intervention Acceptability
Description: Satisfaction with intervention content, delivery, length using a client satisfaction questionnaire and as measured on a likert scale response and as open-ended response options
Time Frame: Acceptability will be assessed during the intervention, an expected average timeframe of 8-14 weeks
Population: Only participants who received intervention were assessed for acceptability through semi-structured interviews
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 0 | 25
Participants |  | 25

5. Secondary Outcome: Number of Participants With Intervention Feasibility
Description: Intervention feasibility measured by attendance, retention for outcome assessments, fidelity
Time Frame: Feasibility will be assessed during the intervention, an expected average timeframe of 8-14 weeks
Population: Only participants randomized to the intervention arm were assessed for feasibility (% of the 41 participants participating in the full intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 0 | 41
Participants | 0 | 37

6. Other Pre Specified Outcome: Time to Event Analysis of ART Initiation
Description: Investigators will perform a Time to Event Analysis of Treatment Initiation and compare this between control and intervention arms.
  Data not available - only measured at 3 months to capture the importance of early treatment initiation
Time Frame: 6 months
Population: No time-to-event analysis carried out
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Number of Participants Who Reported Having Fewer Drinks at 6 Months Than at Baseline
Description: Assessed through self-reported measures of alcohol use: percent reporting fewer daily drinks at six months than at baseline.
  Participants were asked "How often do you have a drink containing alcohol (like beer, wine, or liquor)?" (Never, less than monthly, monthly....4 or more times a week). If they gave an answer other than "Never," they were then asked "How many drinks of any kind containing alcohol do you have on a typical day when you are drinking?" (1 or 2; 3 or 4...10 or more).
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 35 | 29
Participants | 3 | 7

8. Other Pre Specified Outcome: Short-form 8 (SF-8)
Description: Change in self-reported General Health over time. We compared the difference in scores between baseline and six months.
  The SF-8 is an eight question survey for measuring general physical and mental health. It is a shortened version of the SF-36 and the results are interpreted using the same methods. First, items are recorded on a 0 (lowest score) to 100 (highest score) scale, per a scoring key developed by RAND. Then, items in the same scale are averaged together so that each scale representing different elements of health has its own score. Scores represent the average for all questions the participant answered (the percentage of total possible score achieved). The higher the score, the better the participant's health.
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 38
score on a scale | 0.0 (1.0) | -0.1 (1.1)

9. Other Pre Specified Outcome: Change in Self-reported Coping/Ability to Cope Over Time
Description: Brief COPE. We compared the difference in scores between baseline and six months.
  The Brief COPE was developed by Carver, C. S. and provides a condensed version of the full COPE tool which can be modified by choosing only select scales. We used a 2-item scale (both related to alcohol and drug use, min=1, max=4) based on factor analysis results. Higher scores are worse (more use of alcohol/drugs to feel better/get through). We averaged the 2 items to calculate the scale score.
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 37
score on a scale | 1.53 (0.85) | 1.24 (0.57)

10. Other Pre Specified Outcome: Change in Self-reported Belief in ARV Efficacy/Trust in Antiretrovirals Over Time
Description: Perceptions of ARV Therapy Scale, HCSUS. We compared the difference in scores between baseline and six months.
  ARV efficacy was measured using an 8-item scale. For each item, min=1, max=4. Higher scores are better (higher belief in ARV efficacy).
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: Point change on scale
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 37
Point change on scale | 2.93 (0.34) | 3.00 (0.24)

11. Other Pre Specified Outcome: Medical Outcomes Study (MOS) Social Support Survey
Description: Change in self-reported perceived social support over time. We compared the difference in scores between baseline and six months.
  The Social Support Survey contains four subscales (emotional/informational, tangible, affectionate, and positive social interaction) and an overall social support index. A higher score for any of the subscales or the index indicates higher levels of social support. Each subscale score is calculated by finding the average of all the scores in that subscale. The index is found by calculating the average of all the items. Social support was measured by asking eight questions each with a scale of one to five (five being the most support). The minimum score was 8 (least social support) and the maximum was 40 (most social support).
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 37
score on a scale | 4.22 (0.64) | 4.39 (0.65)

12. Other Pre Specified Outcome: Patient-Health Questionnaire (PHQ)-9
Description: Change in self-reported depression over time. We compared the difference in scores between baseline and six months.
  Depression and anxiety symptoms and somatic complaints were measured using the 9-item Patient Health Questionnaire (PHQ), which scores DSM-IV criteria from 0 (not at all) to 3 (nearly every day). The subtotals are summed to create the total score. 0-4 is interpreted as minimal depression, 5-9 as mild depression, 10-14 as moderate depression, 15-19 as moderately severe depression, and 20-27 as severe depression.
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 37
score on a scale | 0.61 (0.56) | 0.32 (0.24)

13. Other Pre Specified Outcome: Change in Self-reported Internalized Stigma Over Time
Description: Internalized Stigma measure developed by Kalichman et al. We compared scores at baseline and six months.
  Internalized stigma was measured using the Internalized AIDS-Related Stigma Scale. This six-item scale is used to measure internalized stigma. Participants either agree (which scores them a "1") or disagree (which scores them a "0") to each item and the total scale score is computed as the sum of the items with a minimum score of 0 and maximum score of 6. The higher the score, the higher their internalized stigma.
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 37
score on a scale | 2.61 (1.50) | 2.30 (1.26)

14. Other Pre Specified Outcome: Change in Self-reported Disclosure Concerns Over Time
Description: Disclosure concerns measure using Berger's HIV Stigma Scale. We modified the instrument to include eight statements related to disclosure concerns (i.e. I regret having told some people that I have HIV; I want to keep my HIV a secret) and participants responded disagree or agree. Disclosure concerns were measured by asking a set of eight questions, with a minimum score of 8 and a maximum score of 16. The higher the score, the greater the level of concern. We compared scores at baseline and six months.
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 37
score on a scale | 3.47 (1.72) | 3.81 (1.61)

15. Other Pre Specified Outcome: Change in Self-reported Anticipated Stigma Over Time
Description: Anticipated Stigma measure developed by Earnshaw et al. We used the HIV Stigma Framework to measure anticipated HIV stigma. This instrument consists of items relating to anticipated stigma from friends, family, and healthcare workers. Items were scored on 5-point Likert-type scales (1=very unlikely, 5=very likely). Higher scores indicate greater anticipated stigma.
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey. In this case, only one participant had not disclosed, but they were determined ineligible for the study.
Time Frame: baseline and 6 months
Population: This scale was only administered to those who had not disclosed HIV status to anyone. Data were collected from 1 participant originally randomized to the intervention arm, but this participant was deemed ineligible.
  The 1 participant who did not report disclosing to anyone chose 2 ("unlikely") for all 9 of the Anticipated Stigma items.
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Change in Self-reported Barriers and Competing Needs Over Time
Description: Barriers and Competing Needs measure developed by Craw JA et al. We compared results at baseline and six months.
  Barriers and competing needs were assessed by asking participants whether they had experienced each of 13 problems when medical care was needed in the past six months (e.g. not knowing where to find care, affordability of medications or transportation). The count of each participant's "yes" responses to these 13 yes/no items was taken as their score. Higher score means more barriers/competing needs.
  Note: 84 participants were enrolled into the study, but not all of them agreed to complete each survey.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Treatment Ambassador Intervention
Number analyzed (Participants) | 43 | 37
score on a scale | 4.55 (2.50) | 3.91 (2.17)

ADVERSE EVENTS:
Time Frame: Six months - the full duration of the study
Arm/Group | Standard of Care | Treatment Ambassador Intervention
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/37
Other Adverse Events (participants affected / at risk) | 0/43 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT03099707/Prot_SAP_000.pdf